CLINICAL TRIAL: NCT04572477
Title: The Influence of Sequential Tau Protein and Amyloid Plaque Imaging Changes on Stroke Prognosis and Cognitive Outcome
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 201601675A0
Record Dates: First submitted 2020-09-29; First posted 2020-10-01 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-04

CONDITIONS: Post-stroke Dementia, Vascular Mild Cognitive Impairment
MeSH Terms: interventions — THK5351; florbetapir

STUDY DESIGN:
Intervention Model Description: Group A (acute stroke/TIA patients), n=200 Group B (chronic stroke/TIA patients), n=200 Group C (healthy elderly controls), n=30
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- [18F]THK-5351 (Other): 1. Primary endpoint A. To compare the distribution of cerebral amyloid plaques and tau protein between stroke patients and normal controls.
  2. Secondary endpoints A. To compare tau distribution on [18F]THK5351 PET at acute, subacute and chronic stroke stages.
  B. To correlate the [18F]THK5351 PET findings with [18F]AV45 PET, brain MRI, and functional and cognitive performance.
  C. To compare the [18F]THK5351PET, [18F]AV45 PET, and brain MRI findings among stroke patients with no cognitive impairment (NCI), storke patients with VaMCI and stroke patients with PSD.
  Interventions: Drug: [18F]THK-5351; Drug: [18F]AV-45
- [18F]AV-45 (Other): 1. Primary endpoint A. To compare the distribution of cerebral amyloid plaques and tau protein between stroke patients and normal controls.
  2. Secondary endpoints A. To compare tau distribution on [18F]THK5351 PET at acute, subacute and chronic stroke stages.
  B. To correlate the [18F]THK5351 PET findings with [18F]AV45 PET, brain MRI, and functional and cognitive performance.
  C. To compare the [18F]THK5351PET, [18F]AV45 PET, and brain MRI findings among stroke patients with no cognitive impairment (NCI), storke patients with VaMCI and stroke patients with PSD.
  Interventions: Drug: [18F]THK-5351; Drug: [18F]AV-45

INTERVENTIONS:
Drug: [18F]THK-5351 — F-18 THK PET Imaging
Drug: [18F]AV-45 — F-18 AV45 PET Imaging

SUMMARY:
Amyloid plaques and tau protein are the landmarks of neurodegeneration in Alzheimer's disease (AD). On the other hand, it is reported that cerebral ischemia may induce amyloid plaques and tau protein accumulation. However, it was difficult to in vivo disentangle the complex and dynamic interactions between AD pathophysiology and cerebral vascular injury in the development of post-stroke cognitive impairment in the past. With the advent of novel radiotracers specific to cerebral amyloid plaques and tau protein, we aim to conduct a prospective multimodal neuroimaging cohort study to investigate the contribution of vascular injury, amyloid plaques and tau protein to stroke recovery and post-stroke cognitive impairment.

ELIGIBILITY:
Inclusion Criteria:

1. Inclusion criteria for acute stroke/TIA patients (Group A, n=200)

   * Males or females with age >= 50 years old
   * Having acute cerebral stroke or transient ischemic attack in recent 1 month
   * Female subjects of childbearing potential must practice effective contraception during the study and be willing and able to continue contraception after the final study
   * Provision of signed informed consent
2. Inclusion criteria for chronic stroke/TIA patients (Group B, n=200)

   * Males or females with age >= 50 years old
   * Having cerebral stroke or transient ischemic attack in the past 1.5 years
   * Having had tau PET imaging study within 1 year after the index stroke/TIA event
   * Female subjects of childbearing potential must practice effective contraception during the study and be willing and able to continue contraception after the final study
   * Provision of signed informed consent
3. Inclusion criteria for healthy elderly controls (Group C, n=30)

   * Males or females with age >= 50 years old
   * Without history of cerebral stroke or transient ischemic attack
   * Ability to participate in cognitive and neuroimaging assessments
   * Female subjects of childbearing potential must practice effective contraception during the study and be willing and able to continue contraception after the final study
   * Provision of signed informed consent

Exclusion Criteria:

Exclusion criteria for all subjects

* Presence of dementia diagnosis before the index stroke or at the initial screening
* History of vascular MCI (VaMCI)
* The Chinese version of the Informant Questionnaire on Cognitive Decline in the Elderly (IQCODE) score >=104 at the initial screening 47.
* Life expectancy less than 1 year.
* Clinically significant abnormal laboratory values.
* Clinically significant or unstable medical or psychiatric illness.
* Epilepsy history.
* Cognitive impairment resulting from trauma or brain damage.
* Substance abuse or alcoholism in the past 3 months.
* General MRI, and / or PET exclusion criteria.
* Pregnant or becoming pregnant during the study (as documented by pregnancy testing at screening or at any date during the study according to the PI discretion) or current breast feeding.
* History of allergy to 18F-labelled radionucleic agents, [18F]AV45 or [18F]THK5351.
* Subjects having high risks for the study according to the PI discretion.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2017-06-01 (Actual); Primary Completion 2023-11-30 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
Imaging positive and negative conditions | through study completion, an average of 1.5 year
  PET images are visually assessed by independent raters, who are nuclear medicine doctors and blinded to all clinical and diagnostic information. The raters classify each scan as 0-1 (no significant uptake)、2 (suspicious uptake)、3-4 (significant uptake). The score >= 2 is deemed as positive condition.
Chi-square test will be performed to analyze dementia conversion rate. | through study completion, an average of 1.5 year

CONTACTS AND LOCATIONS:
Overall Officials: Huang Kuo-Lun, M.D., Study Chair — Stroke Section, Department of Neurology, Chang-Gung memorial Hospital
Locations (1):
- Department of Neurology, Chang-Gung memorial Hospital, Taoyuan District, Guishan, Taiwan